CLINICAL TRIAL: NCT06711731
Title: The Freiburg Registry on SpontanEous IntercrAnial Hypotension (SIH) & Post-duraL Puncture Headache (PDPH)
Acronym: SEAL
Status: Recruiting | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Myriam Peters, Scientist, University Hospital Freiburg
Other Study IDs: 24-1357-S1
Record Dates: First submitted 2024-11-15; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: CerebroSpinal Fluid (CSF) Leak
Keywords: SIH; PDPH; Spinal leaks; CSF leak; SLEC; Spontaneouse Intercranial Hypotension; CSF-venous fistula; Post Dural Puncture Headache; Cerebrospinal Fluid Leak; Rare disease
MeSH Terms: conditions — Cerebrospinal Fluid Otorrhea; Post-Dural Puncture Headache; Cerebrospinal Fluid Leak; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- spinal CSF leak: Patients with suspected spinal CSF leak based on one of the following:
  1. History of new orthostatic symptoms with or without prior spinal procedure
  2. Imaging suggestive for spinal CSF leak

SUMMARY:
Spinal CSF leaks are considered as rare disease. They cause a variety of symptoms, mainly culminating in a chronic headache syndrome. Crucially, yet often disregarded, the disease holds the potential for cure. The multitude of symptoms, and their inconsistency over time are just two of many challenges preventing timely diagnosis and treatment in many patients.

Spinal CSF leaks can occur after intentional or accidental dural puncture (post-dural puncture headache - PDPH) or spontaneously (spontaneous intracranial hypotension - SIH). Awareness is steadily increasing with simultaneous increase of recognized patients. Yet, research and diagnostic is mainly provided by few specialized centers, as e.g. Freiburg. Thus, many observations point towards a large non-diagnosed and non-recognized number of patients, most likely being misdiagnosed and mistreated.

Objective: The aim of the registry is to collect structured information on the frequency, cause, symptoms, diagnostic procedures, treatment options and long-term outcome. With the help of the registry, we would like to contribute to a better understanding and treatment of the diseases.

Methods: Prospective, longitudinal registry on patients with suspected SIH or PDPH, including data on demographics, clinical presentation, diagnostic findings, treatment, at treatment outcome.

DETAILED DESCRIPTION:
Spinal CSF leaks have a severe impact on quality of life and health. Symptoms vary from chronic headache syndrome to intracranial bleeding, cognitive decline, and coma. Crucially, yet often disregarded, the disease holds the potential for cure.

Lumbar dural leaks can arise from commonly performed medical interventions such as diagnostic lumbar punctures, spinal anesthesia, spinal infiltrations, or incidental dural punctures during epidural analgesia in obstetric care, resulting in post-dural puncture headache (PDPH).

Additionally, a notable fraction of spinal CSF leaks manifests as spontaneous intracranial hypotension (SIH), which derives from different types of spontaneous leaks along the Spine and remains broadly under-recognized.

The main clinical symptoms of spinal CSF leaks are orthostatic headaches with a most often defined beginning, typically accompanied by hearing impairment and dizziness, worsened by exercise and movement. Additionally, other manifestations are known, such as cognitive decline, bilateral brachial amyotrophy, paradox headache, fatigue, and many more. In patients presenting with spinal CSF leaks, the accurate diagnosis often eludes clinicians, leading to frequent misdiagnoses of chronic migraine, fatigue, or psychiatric conditions. Many patients endure months, if not years, before a diagnosis of a treatable condition is finally established. The heterogeneity of the symptoms can appear inconsistent or even paradoxical, posing diagnostic challenges. The extent of possible long-term deterioration is not recognized.

The reported incidence of PDPH fluctuates considerably, ranging from 2 to 40 per 100 procedures performed. This variance is influenced by patient-related factors (e.g., age, gender, pregnancy status) and procedural factors (e.g., needle size and type). PDPH, according to current criteria, occurs within 5 days after a dural puncture. Nevertheless, there are widely underestimated pitfalls: a dural puncture is not always recognized by the person performing an epidural procedure, symptoms can occur after more than 5 days, and disease courses can be chronic. These facts are widely unknown, leading to largely hidden figures of patients being under or misdiagnosed and, thus, not treated. Moreover, PDPH is primarily observed following unintentional dural puncture during the administration of obstetric anaesthesia and analgesia to parturients.

Spontaneous intracranial hypotension (SIH) can be caused by ventral, lateral, or sacral spinal leaks or by CSF-venous fistulae, which was first described in 2014. An annual incidence rate of ~ 4/100,000 was estimated in 2022. This rate is likely underestimated as it only includes confirmed cases, thus recognized cases within a widely non-recognized entity. Often, patients are neither identified nor directed to the appropriate MRI, which, in numerous instances, could lead to the correct diagnosis. Even when SIH is identified, non-targeted epidural blood patches in the lumbar region are often not administered due to perceived elevated risks. An epidural blood patch might be able to help to heal the leak. At the same time, it must be noted that even long-term improvement does not necessarily indicate closure of the leak and prevention of long-term sequelae, such as superficial siderosis. Invasive diagnostics are not employed to pinpoint the location, and treatment to seal the leak is not consistently pursued. The effects of treatment are often immediate and can be successful even in chronic patients. Evidence shows that leaks are held open by new membranes (Neo-membranes) that prevent spontaneous healing. Thus, the correct localization of such a leak and targeted sealing or close follow-ups should be initiated.

The management approaches for SIH and PDPH significantly deviate from standard pain management strategies employed for other types of headaches. Noteworthy interventions include the application of blood patches and even surgical measures to seal the leak, offering curative solutions. Those enduring chronic spinal CSF leaks experience profound limitations in their health-related quality of life, comparable to those with chronic immunological diseases or cancer. Overlooking the diagnosis and management of spinal CSF leaks may precipitate progressive deterioration, with the potential for persistent sequelae like superficial siderosis, syndromes mimicking frontotemporal dementia (FTD), and chronic subdural hematoma formation.

This registry aims to set ground for standardized, prospective demographic, diagnostic and treatment data assessments, and patient self-reported outcome measures.

Collecting this data is essential to potentially exploring risk factors, understanding outcome predictors, and refining diagnostics. Additionally, standardized data collection will allow the appropriate designing of urgently needed randomized trials.

Aims:

Primary aim:

To describe the proportion of patients diagnosed with SIH or PDPH

Secondary aims:

1. To describe the proportion of different spinal CSF leaks observed per entity
2. To describe the demographics per entity, and per different spinal CSF leak type
3. To describe the clinical spectrum per entity, and per different spinal CSF leak type
4. To describe the imaging features per entity, and per different spinal CSF leak type
5. To describe the outcome of different treatments, and per different spinal CSF leak type
6. To describe the adverse events of different treatments, and per different spinal CSF leak type
7. To explore potential diagnostic markers per entity, and per different spinal CSF leak type
8. To explore risk factors per entity, and per different spinal CSF leak type
9. To evaluate differences between spinal CSF leak types regarding age, sex, BMI, clinical presentation, diagnostic findings
10. To assess the effect of disease duration on imaging findings, and on outcome after persistent closure of a leak

Method:

The registry is prospective, longitudinal and currently monocentric*. Diagnostic, treatment, and follow-up procedures follow clinical standard operating procedures (SOP) according to the suspected diagnosis and the clinical findings.

Routinely assessed data of the initial diagnostic workup and the individual's disease course with or without treatment will be collected over 2 years per individual. The investigators' semi-annual meetings ensure the achievement of the register's predefined aims.

There are no specific risks or benefits for the patients participating in this registry. Any procedure will be performed according to clinical standards as indicated. There will be no additional visits to the hospital or the ambulatory. There will be no additional imaging performed, especially no additional radiation.

A merely intrinsic benefit might exist for the patient supporting this study and supporting medical research.

As this is an explorative and observational study on rare diseases without formal sample size estimation, we limit the study by time of duration (10 years).

Patients suffering from rare diseases most often face delays in diagnostics and treatments. To underscore this known burden: By an estimated population of 1.74 Mio in the Freiburg area and an incidence rate of SIH of about 5/100.0004, approximately 85 patients should be expected per year stemming from this area. Freiburg is the only center offering adequate diagnostic pipelines for these patients. Despite the increasing awareness, the number of patients diagnosed in the area adjunct to the Freiburg CSF center is within a range of 15 to 20 patients per year, thus still too low compared to the expected number with many patients unrecognized, and or underdiagnosed.

Our current numbers of confirmed SIH treatments range from 100 per year with patients being referred throughout Germany and about 15-20 international patients per year. We expect this rate to rise within the next few years. The number of PDPH patients with a focus on persistent PDPH patients is currently rapidly increasing. We see about 40-60 per year.

Interim-Evaluation of the Registry's primary and secondary descriptive aims will be performed and reported as a step-wise, dynamic approach:

* After each +100 patients with confirmed SIH
* After each +50 patients with confirmed PDPH

The secondary objectives, which involve comparisons, the exploration of diagnostic markers, and risk factors, will be addressed using a dynamic biostatistical model: The analysis will only be conducted after a power analysis deems the observed sample adequate.

Proportions will be presented as a percentage with 95% confidence interval (CI).

The sata of patients with different types of spinal CSF leaks will be summarized using descriptive statistics, i.e. median and quartiles for continuous and absolute and relative frequencies for categorical variables, regarding their clinical, laboratory, and diagnostic findings, and number of diagnostic and therapeutic procedures needed.

Furthermore, the proportion of SIH patients with different spinal CSF leak types

1. will be compared between males and females using a Chi2-Test and a risk difference with 95% CI.
2. Will be presented by age groups (per two decades), and per sex as a percentage with a 95% Wilson confidence interval (CI).

Age, sex, BMI, clinical presentation, and diagnostic findings between different spinal CSF leaks will be compared using the Mann-Whitney-Wilcoxon test and Chi2 test for continuous and categorical variables, respectively.

A multivariable logistic regression for the presence of SIH, PDPH, and chronic PDPH, respectively, will be constructed using the clinical and diagnostic parameters with some evidence for a difference according to the presence of a spinal CSF leak (p < 0.2). The potential nonlinearity of the age effect is evaluated based on a residual analysis of the regression model. Odds ratios with 95% CI will be reported. Using bootstrapping, we will present a ROC curve and AUC with 95% Due to the exploratory approach,, no correction for multiple testing will be performed.

A multivariable linear regression for imaging findings (especially Bern Score, presence of SLEC, vand olumetries), and for the patient-reported outcomes will be constructed using the clinical and diagnostic parameters at admission with some evidence for a difference (p<0.2). Adjusted R-squares, Beta-coefficients with 95% CI, standard errors will be reported.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected spinal CSF leak based on one of the following

   * History of new orthostatic symptomes with or without prior spinal procedure
   * Imaging suggestive for spinal CSF leak
2. Informed consent

Exclusion Criteria:

a) Symptoms beeing conclusively explained by another known diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The registry is an explorative study on patients suffering from a rare disease - therefor it is aimed to include all eligible patients for a time-limit of 10 years. All patients with suspected spinal CSF leak will be approached and informed about the registry. In case of legal incapacity, the caregivers will be approached. The inclusion of this vulnerable group is considerable as they represent a small but very important subgroup of patients suffering from demntia stemming from a traetable cause.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2034-12-04 (Estimated); Study Completion 2036-12-04 (Estimated)

PRIMARY OUTCOMES:
Primary Diagnosis given after primary workup (yes/no) | up to 4 weeks after inclusion
  * SIH (fulfilling ICHD-3 criteria) - yes/no
  * atypical SIH - yes/on
  * Asymptomatic SIH (positive imaging signs only) - yes/no
  * PDPH (fulfilling ICHD-3-criteria) - yes/no
  * persistentPDPH - yes/no

SECONDARY OUTCOMES:
SIH/PDPH - Experience of the local team | at time of inclusion
  Number of patient with suspicion for SIH work-up/year
SIH/PDPH - Patients' demographics | at time of inclusion
  Country, City
SIH - Previously received treatment at time of inclusion (yes/no) | at time of inclusion
  Medical SIH treatment, Other symptomatic treatment, Untargeted lumbar blood patch, Targeted blood patch, Targeted fibrin patch, Endovascular embolization, Minimally invasive surgery, Open surgery - dorsal approach, Open surgery-ventral approach, Open surgery-transforaminal approach, Discectomy, Laminectomy, Stabilization procedures, Surgery, other techniques
SIH/PDPH - age | at time of inclusion
  years
SIH/PDPH - sex | at time of inclusion
  male female diverse
SIH/PDPH - height | at time of inclusion
  height in meter (m)
SIH/PDPH - weight | at time of inclusion
  kilogram (kg)
SIH/PDPH - modified Ranking scale | at time of inclusion
  range in 0-6, 0 indicating best health
SIH/PDPH - pre-existing Neurological deficits (yes/no) | at time of inclusion
  Neurological deficits due to previously attempted treatments at the time of inclusion
SIH/PDPH - Neurological deficits in routine clinical testing | at time of inclusion
  descriptive
SIH - Montreal cognitive Assessment | at time of inclusion
  range 0-30, 30 indicating best performance
SIH - Trail-making test part B | at time of inclusion
  in minutes needed to fulfill the task
PDPH -BMI | at time of inclusion
  kg/m^2
SIH/PDPH - Regular use of stimuli > 6 months (yes/no) | at time of inclusion
  Nicotine, Alcohol, Recreational drugs
SIH/PDPH - Headache-Impact-Test (HIT)-6 | at time of inclusion
  Headache-Impact-Test (HIT)-6 range 36 to 78 points, 78 indicating highest impact of headaches.
SIH/PDPH - 5 dimensions /5 levels European Quality of life questionaire (EQ-5D-5L) Index | at time of inclusion
  <0 to 1, with 1 indicating unimpaired health
SIH/PDPH - Self-Administered Comorbidity Questionaire (SCQ) | at time of inclusion
  13-item Self-Adminestered Comorbidity Questionaire (SCQ), range 0 to 39, 0 indicating lowest burden
PDPH - Patient'S Global Impression of Change (PIGC) | at time of inclusion
  range 7 - 42, 7 indicating highest improvement
SIH - Opening pressure on lumbar puncture if performed (not recommended in routine), or myelogram | up to 4 weeks
  cmH2O
SIH/PDPH - Total Bern-Score MRI head according to Dobrocky et al. | up to 4 weeks
  range 0 to 9 with 9 indicating highest likelihood of a spinal CSF leak
SIH/PDPH - Subitems Bern-Score MRI head according to Dobrocky et al. | up to 4 weeks
  Meningeal enhancement (yes/no), Subdural fluid (yes/no), Venous Distention (yes/no), Effaced suprasellar distance (yes/no), Effaced mamillopontine distance (yes/no), Effaced prepontine distance (yes/no)
SIH - MRI head - Superficial Siderosis | up to 4 weeks
  (yes/no)
SIH - MRI head - Layered calvarial hyperostosis | up to 4 weeks
  (yes/no)
SIH - Sinus vein thrombosis | up to 4 weeks
  (yes/no)
SIH/PDPH - Volumetry of the CSF-space MRI head & spine | up to 4 weeks
  mm^3
SIH/PDPH - Volumetry of the CNS MRI head & spine | up to 4 weeks
  mm^3
SIH/PDPH - Imaging Density score | up to 4 weeks
  Density scores of the intracranial compartments MRI head & spine
SIH/PDPH - Total radiation dose applied per diagnostic procedure with radiation performed | at primary workup
  Sievert
SIH - Myelography number | up to 24 weeks
  Number of myelographies performed for precise localization
SIH - Type of myelography technique applied (yes/no) | up to 4 weeks
  conventional,digital subtraction, dynamic CT, Cone-beam CT, Photon-counting CT, fluoroscopy, Other (specify)
SIH - Adverse events during myelography (yes/no) | up to 4 weeks
  nausea, dizziness/vertigo, emesis, allergic reaction, seizure, treatment intensive care unit (independent of cause))
SIH - Headache before and after myelogram | up to 4 weeks
  in 0-10, 10 numeric rating scale
SIH - Positioning during index myelography that proofs the leak (yes/no) | up to 4 weeks
  prone, lateral decubitus, supine
SIH - myelography that proofs the leak performed applying (yes/no) | up to 4 weeks
  resisted insipration, pressuization, valsalva maneuver
SIH/PDPH - Lumbar Infusiontest - Pressure at baseline | up to 4 weeks
  pressure (mmHg)
SIH/PDPH - Lumbar Infusiontest - Resistence to CSF outflow (Rcsf) | up to 4 Weeks
  mmHg/(ml/min)
SIH/PDPH - Lumbar Infusiontest - Elastance | up to 4 weeks
  Elastance coefficient (1/ml)
SIH/PDPH - Lumbar Infusiontest - Pressure-Volume-Index | up to 4 weeks
  ml
SIH/PDPH - Lumbar Infusiontest - Needle resistance | up to 4 weeks
SIH/PDPH - PET-CT - Evidence of CSF-loss (yes/no) | up to 4 weeks
SIH/PDPH - PET-CT if performed - | up tp 4 weeks
  half-life of the tracer in the CSF space (minutes)
SIH/PDPH - Laboratory parameters at diagnosis (normal/abnormal) | up to 4 weeks after inclusion
  * complete routine Blood analysis (including: cellcount, electrolytes, coagulation, renal function, thyroid marker) (normal/abnormal)
  * complete routine CSF-analysis (including: cell count, protein) (normal/abnormal)
SIH - CSF leak types identified by dynamic myelography (yes/no) | up to 4 weeks
  * Ventral dural leak
  * Lateral dural leak
  * CSF-venous fistula, single
  * CSF-venous fistula, multiple
  * Sacral dural leak
  * CSF-lymphatic fistula
  * Dorsal dural leak
  * Undefined
SIH - Multiples leaks (yes/no) | up to 4 weeks
SIH - Level of spinal CSF leak (spinal segment) and side in myelogram | up to 4 weeks
SIH - In case of surgery: spinal segment and side confirmed? (yes/no) | up to 4 weeks
SIH/PDPH - Experience of leading interventionalist in SIH-diagnostics/year | up to 4 weeks
SIH/PDPH - Disease duration at time of therapy | up to 4 weeks
  month
SIH/PDPH - Therapy performed after CSF leak diagnosis (yes/no) | up to 4 weeks
  Untargeted lumbar blood patch, Targeted blood patch, Targeted fibrin patch, Endovascular embolization, Minimally invasive surgery with patching, Minimally invasive surgery with clipping, Minimally invasive surgery with disconnection, Open surgery, dorsal approach, Open surgery, ventral approach, Open surgery, transforaminal approach, Surgery, other techniques, Medical PDPH treatment, Other symptomatic treatment, e.g. infiltration N. occipitalis, Untargeted lumbar platelet-rich fibrin patch
SIH/PDPH - Experience of leading surgeon in SIH/PDPH-surgeries/year | up to 4 weeks or longer, depending on the number of surgeries
  in numbers of SIH/PDPH-surgeries/year
SIH/PDPH - Interventions needed addressing secondary complications of spinal CSF leaks, especially chronic subdural hematoma | up to 4 weeks
  Twist drill craniostomy (yes/no), Burr hole craniostomy (yes/no ), Mini craniotomy (yes/no), Conventional trepanation (yes/no), Use of drains and any form of controlled lavage (saline and or clot lysis) (yes/no,), Embolization of MMA (middle meningeal arteria) (yes/no), Other intervention (yes/no)
PDPH - Event of putative dural puncture | up to 4 weeks
  date
PDPH - Event of putative dural puncture (yes/ no) | up to 4 weeks
  * Diagnostic lumbar puncture
  * Diagnostic lumbar puncture with drainage in idiopathic intracranial hypertension
  * Diagnostic lumbar puncture with drainage in idiopathic normal-pressure hydrocephalus
  * Peridural anesthesia in obstetrics
  * Spinal anesthesia in obstetrics
  * Peridural anesthesia, other intervention
  * Spinal anesthesia, other intervention
  * Infiltration
  * others
SIH/PDPH - adverse events related to current treatment at discharge (yes/no) | up to 4 weeks
  Rebound hypertension, Persistence/Reoccurrence of the leak, Suture insufficiency, Infect (systemic/local), Bleeding, Sensory deficits, Motor deficits, Gait ataxia, Bladder dysfunction, Bowl dysfunction, Others
PDPH - Lumbar segment of putative dural puncture known (yes/no) | up to 4 weeks
PDPH - Puncture under imaging guidance | up to 4 weeks
  "location truly known"
PDPH - Duration between (putative) dural puncture until the onset of symptoms | up to 4 weeks
  days
PDPH - Time to first blood patch | up to 4 weeks
  days
PDPH - Number of bloodpatches received before admission | up to 4 weeks
PDPH - Prior treatments at the time of admission (yes/no) | up to 4 weeks
  Fluids, Caffeine, Bedrest, Medical treatment, Other treatment, e.g., infiltrations, Untargeted lumbar bloodpatch, Surgery
PDPH - Post-dural puncture pseudomeningocele ("arachnoid bleb") | up to 4 weeks
  (yes/no)
PDPH - Spinal Segment location of the "arachnoid bleb" | up to 4 weeks
PDPH - Identified CSF leak types by dynamics myelography and/or intraoperatively: | up to 4 weeks
  ventral post-dural puncture leak, dorsal post-dural puncture pseudomeningocele ("arachnoid bleb"), dorsal post-dural puncture leak None
PDPH - Intraoperatively Identified membranes (yes/no) | up to 4 weeks
  neo-membranes (pseudo dura), webs, funnels
PDPH - Dinosaur-tail sign (yes/no) | at time of inclusion
PDPH - specific segment of identified intraoperative membranes (descriptive) | up to 4 weeks
PDPH - CSF leak types identified by dynamic myelography and/or intraoperatively | up to 4 weeks
  ventral post-dural puncture leak, dorsal post-dural puncture pseudomeningocele ("arachnoid bleb"), dorsal post-dural puncture leak, None
PDPH - Diagnostic procedures performed (yes/no, number) | uo to 4 weeks
  CT Head, MRI head, MRI spine, Dynamic digital subtraction myelogram, Dynamic CT-myelogram, Photon-counting CT-myelogram, Cone-beam myelogram, Infusion testing, PET-CT, Other (to exclude/confirm alternative diagnosis)
PDPH - Volume lumbar bloodpatch | up to 4 weeks
  ml
SIH/PDPH - work capacity | at time of inclusion
  range 0 to 5, 0 indicating full capacity
SIH/PDPH -complaints | at time of inclusion
  * current complaints (descriptively)
  * most stressful complaint (descriptively)
SIH/PDPH - headache severity | at time of inclusion
  range 0 to 10, 10 indicating most severe pain
SIH/PDPH - Days within the last month | at time of inclusion
  * with headaches
  * with pain medication intake in the last month
SIH/PDPH - maximum duration being continuously upright | at time of inclusion
  hours
SIH/PDPH - severeness of dizziness | at time of inclusion
  - in 0 to 10, 10 being most severe
SIH/PDPH - Severeness of shoulder- and neck pain | at time of inclusion
  - in 0 to 10, 10 being most severe
SIH/PDPH - severeness of nausea | at time of inclusion
  - in 0 to 10, 10 being most severe
SIH/PDPH - severeness of hearing disturbances and tinnitus | at time of inclusion
  - in 0 to 10, 10 being most severe
SIH/PDPH - severeness of cognitive deficits | at time of inclusion
  - in 0 to 10, 10 being most severe
SIH/PDPH - severeness of visual disturbances | at time of inclusion
  - in 0 to 10, 10 being most severe
SIH/PDPH - . ability to focus and concentrate | at time of inclusion
  rated between 0 to 5, with 5 indicating highest burden
SIH/PDPH - MRI spine: Spinal longitudinal extradural fluid collection (SLEC) (yes/no) | up to 4 weeks
SIH/PDPH - MRI-spine: DiverTICula (TIC) ≥8mm (yes/no) | up to 4 weeks
  number of TICs ≥8mm
SIH/PDPH - Volumetry of epidural spinal veins at C2 | up to 4 weeks
  mm^3
SIH/PDPH - MRI spine: Enlarged cervical epidural spinal veins at C2 | up to 4 weeks
  yes/no
SIH/PDPH - lumbar infusion test - pressure at tilt down | up to 4 weeks after inclusion
  mmHg
SIH/PDPH - lumbar infusion test - pressure at tilt up 10° | up to 4 weeks after inclusion
  mmHg
SIH/PDPH - lumbar infusion test - pressure at tilt up 30° | up to 4 weeks after inclusion
  mmHg
SIH/PDPH - lumbar infusion test - pressure at plateau | up to 4 weeks after inclusion
  mmHg
SIH/PDPH - Laboratory parameters at diagnosis (decriptive) | up to 4 weeks after inclusion
  * Routine Blood analysis
  * Abnormal CSF-analysis
SIH/PDPH - Lumbar Infusiontest - amplitude at baseline | up to 4 weeks
  mmHg
SIH/PDPH - lumbar infusion test - amplitude at tilt down | up to 4 weeks after inclusion
  mmHg
SIH/PDPH - lumbar infusion test -amplitude at tilt up 10° | up to 4 weeks after inclusion
  mmHg
SIH/PDPH - lumbar infusion test - amplitude at tilt up 30° | up to 4 weeks after inclusion
  mmHg
SIH/PDPH - lumbar infusion test - amplitude at plateau | up to 4 weeks after inclusion
  mmHg
SIH/PDPH - PET-CT if performed - | up tp 4 weeks
  half-life of the tracer o0ver the convexities (minutes)
SIH/PDPH - Results of neuropathological tissue analysis if assessed (descriptive) | up to 6 weeks
  epidural membranes (descriptive) arachnoid funnels (descriptive) diverticula (descriptive) epidural vessels (descriptive)
SIH/PDPH - phase-contrast MRI : CSF-velocity | up to 4 weeks
  cm/s
SIH/PDPH - phase-contrast MRI: Stroke-volume CSF | up to 4 weeks
  ml
SIH/PDPH - phase-contrast MRI: Spinal cord motion | up to 4 weeks
  mm
SIH/PDPH - phase-contrast MRI: Spinal cord velocities | up to 4 weeks
  cm/s
SIH/PDPH - MRI spine: Bud-on-branching sign (yes/no) | up to 4 weeks
SIH/PDPH - MRI spine: Localized flow-voids in sagittal spine T2 images (yes/no) | up to 4 weeks

OTHER OUTCOMES:
SIH/PDPH - Follow up-Reported adverse events related to treatment (yes/no) | 4 weeks and 3 month after treatment
  Rebound hypertension, Reoccurrence of the leak, Suture insufficiency, Bleeding, Sensory deficits, Motor deficits, Gait ataxia, Bladder dysfunction, Bowl dysfunction, Others
SIH/PDPH - Follow up-Duration of treatment for rebound hypertension after therapy of the CSF leak | 4 weeks after treatment
  days
SIH/PDPH - Follow up-Average dosage of acetazolamide per day | 4 weeks after treatment
  mean mg/d
SIH/PDPH - Follow up - Total Bern-Score, according to Dobrocky et al. | 3 months after treatment
  range 0 to 9, 9 indicating highest likelihood of spinal CSF leak
SIH/PDPH - Follow up - Subitems Bern-Score, according to Dobrocky et al. | 3 months after treatment
  * Meningeal enhancement (yes/no)
  * Subdural fluid (yes/no)
  * Venous distention (yes/no)
  * Effaced suprasellar distance (yes/no)
  * Effaced mamillopontine distance (yes/no)
  * Effaced prepontine distance (yes/no)
SIH/PDPH - Follow up - Spinal longitudinal extradural fluid collection at site of the leak (SLEC) (only if present before) | 3 months after treatment
  yes /no
SIH/PDPH - Follow up - Headache-Impact-Test (HIT)-6 | 3, 6, 12 & 24 months after treatment
  range 36 to 78 points, 78 indicating highest impact of headaches
SIH/PDPH - Follow up - 5 dimension/ 5 levels European Quality of life questionnaire (EQ-5D-5L) | 3, 6, 12, & 24 months after treatment
  <0 to1, 1indicating unimpaired health
SIH/PDPH - Follow up - Patient's Global Impression of Change (PGIC) | 3, 6, 12 & 24 months after treatment
  range 7 to 42, 7 indicating highest improvement
SIH/ PDPH - Follow up - Self-administered comorbidity questionnaire (SCQ) | 12 & 24 months after treatment
  range 0 to 39, 0 indicating lowest burden
SIH/PDPH - follow-up - current working capacity | at 4 weeks & 3, 6, 12 & 24 months
  range 0 to 5, 0 indicating full capacity
SIH/PDPH - follow-up - complaints | 4 week, 3, 6, 12 & 24 months
  * current complaints (descriptively)
  * most stressful complaint (descriptively)
SIH/PDPH - follow-up - headache severity | 4 week, 3, 6, 12 & 24 months
  range 0 to 10, 10 indicating most severe pain
SIH/PDPH - follow-up - Days within the last month | 4 weeks, 3, 6, 12, 24 months
  with headaches with pain medication intake in the last month
SIH/PDPH - follow-up - maximum duration being continuously upright | 4 weeks, 3, 6, 12 & 24 months
  hours
SIH/PDPH - follow-up - severeness of dizziness | 4 weeks, 3, 6, 12 &24 months
  - in 0 to 10, 10 being most severe
SIH/PDPH - follow-up - Severeness of shoulder- and neck pain | 4 weeks, 3, 6, 12 & 24 months
  in 0 to 10, 10 being most severe
SIH/PDPH - follow-up - severeness of nausea | 4 weeks, 3, 6, 12 & 24 months
  in 0 to 10, 10 being most severe
SIH/PDPH - follow-up - severeness of hearing disturbances and tinnitus | 4 weeks, 3, 6, 12 & 24 months
  in 0 to 10, 10 being most severe
SIH/PDPH - follow-up - severeness of cognitive deficits | 4 weeks, 3, 6, 12 & 24 months
  in 0 to 10, 10 being most severe
SIH/PDPH - follow-up - severeness of visual disturbances | 4 weeks, 3, 6, 12 & 24 months
  in 0 to 10, 10 being most severe
SIH/PDPH - follow-up - exhaustion | 4 weeks, 3, 6,12 &24 months
  rated between 0 to 5, with 5 indicating highest burden
SIH/PDPH - follow-up - ability to focus and concentrate | 4 weeks, 3, 6, 12 & 24 months
  rated between 0 to 5, with 5 indicating highest burden
SIH/PDPH - follow-up - phase-contrast MRI: CSF-velocity (if performed) | up to 6 months after treatment
  cm/s
SIH/PDPH - follow-up - phase-contrast MRI Stroke-volume CSF (if performed) | up to 6 months after treatment
  ml
SIH/PDPH - follow-up - phase-contrast MRI Spinal cord motion (if performed) | up to 6 months after treatment
  mm
SIH/PDPH - follow-up - phase-contrast MRI Spinal cord velocity (if performed) | up to 6 months after treatment
  cm/s

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center - University of Freiburg, Germany, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schievink WI, Maya MM, Moser FG, Simon P, Nuno M. Incidence of spontaneous intracranial hypotension in a community: Beverly Hills, California, 2006-2020. Cephalalgia. 2022 Apr;42(4-5):312-316. doi: 10.1177/03331024211048510. Epub 2021 Sep 23. PMID 34553617
- [Background] Lashkarivand A, Eide PK. Brain Sagging Dementia-Diagnosis, Treatment, and Outcome: A Review. Neurology. 2022 May 10;98(19):798-805. doi: 10.1212/WNL.0000000000200511. Epub 2022 Mar 25. PMID 35338080
- [Background] Schievink WI, Maya M, Barnard Z, Tache RB, Prasad RS, Wadhwa VS, Moser FG, Nuno M. The reversible impairment of behavioral variant frontotemporal brain sagging syndrome: Challenges and opportunities. Alzheimers Dement (N Y). 2022 Dec 18;8(1):e12367. doi: 10.1002/trc2.12367. eCollection 2022. PMID 36544987
- [Background] Schievink WI, Maya MM, Harris J, Galvan J, Tache RB, Nuno M. Infratentorial Superficial Siderosis and Spontaneous Intracranial Hypotension. Ann Neurol. 2023 Jan;93(1):64-75. doi: 10.1002/ana.26521. Epub 2022 Oct 22. PMID 36200700
- [Background] Sprave T, Gkika E, Verma V, Grosu AL, Stoian R. Patient reported outcomes based on EQ-5D-5L questionnaires in head and neck cancer patients: a real-world study. BMC Cancer. 2022 Nov 29;22(1):1236. doi: 10.1186/s12885-022-10346-4. PMID 36447175
- [Background] Cella D, Grunwald V, Escudier B, Hammers HJ, George S, Nathan P, Grimm MO, Rini BI, Doan J, Ivanescu C, Paty J, Mekan S, Motzer RJ. Patient-reported outcomes of patients with advanced renal cell carcinoma treated with nivolumab plus ipilimumab versus sunitinib (CheckMate 214): a randomised, phase 3 trial. Lancet Oncol. 2019 Feb;20(2):297-310. doi: 10.1016/S1470-2045(18)30778-2. Epub 2019 Jan 15. PMID 30658932
- [Background] Niraj G, Mushambi M, Gauthama P, Patil A, Kelkar A, Hart E, Nurmikko T; Accidental Dural Puncture Outcome Study Collaborative Group. Persistent headache and low back pain after accidental dural puncture in the obstetric population: a prospective, observational, multicentre cohort study. Anaesthesia. 2021 Aug;76(8):1068-1076. doi: 10.1111/anae.15491. Epub 2021 Apr 23. PMID 33891312
- [Background] Ranganathan P, Golfeiz C, Phelps AL, Singh S, Shnol H, Paul N, Attaallah AF, Vallejo MC. Chronic headache and backache are long-term sequelae of unintentional dural puncture in the obstetric population. J Clin Anesth. 2015 May;27(3):201-6. doi: 10.1016/j.jclinane.2014.07.008. Epub 2014 Dec 4. PMID 25483233
- [Background] MacArthur C, Lewis M, Knox EG. Accidental dural puncture in obstetric patients and long term symptoms. BMJ. 1993 Apr 3;306(6882):883-5. doi: 10.1136/bmj.306.6882.883. PMID 8490410
- [Background] Piechowiak EI, Aeschimann B, Hani L, Kaesmacher J, Mordasini P, Jesse CM, Schankin CJ, Raabe A, Schar RT, Gralla J, Beck J, Dobrocky T. Epidural Blood Patching in Spontaneous Intracranial Hypotension-Do we Really Seal the Leak? Clin Neuroradiol. 2023 Mar;33(1):211-218. doi: 10.1007/s00062-022-01205-7. Epub 2022 Aug 26. PMID 36028627
- [Background] Beck J, Hubbe U, Klingler JH, Roelz R, Kraus LM, Volz F, Lutzen N, Urbach H, Kieselbach K, Fung C. Minimally invasive surgery for spinal cerebrospinal fluid leaks in spontaneous intracranial hypotension. J Neurosurg Spine. 2022 Sep 9;38(1):147-152. doi: 10.3171/2022.7.SPINE2252. Print 2023 Jan 1. PMID 36087332
- [Background] Carlton Jones L, Butteriss D, Scoffings D. Spontaneous intracranial hypotension: the role of radiology in diagnosis and management. Clin Radiol. 2022 Mar;77(3):e181-e194. doi: 10.1016/j.crad.2021.11.007. Epub 2021 Dec 20. PMID 34949452
- [Background] Dobrocky T, Grunder L, Breiding PS, Branca M, Limacher A, Mosimann PJ, Mordasini P, Zibold F, Haeni L, Jesse CM, Fung C, Raabe A, Ulrich CT, Gralla J, Beck J, Piechowiak EI. Assessing Spinal Cerebrospinal Fluid Leaks in Spontaneous Intracranial Hypotension With a Scoring System Based on Brain Magnetic Resonance Imaging Findings. JAMA Neurol. 2019 May 1;76(5):580-587. doi: 10.1001/jamaneurol.2018.4921. PMID 30776059
- [Background] Pradeep A, Madhavan AA, Brinjikji W, Cutsforth-Gregory JK. Incidence of spontaneous intracranial hypotension in Olmsted County, Minnesota: 2019-2021. Interv Neuroradiol. 2025 Jun;31(3):364-368. doi: 10.1177/15910199231165429. Epub 2023 Mar 22. PMID 36945844
- [Background] Farb RI, Nicholson PJ, Peng PW, Massicotte EM, Lay C, Krings T, terBrugge KG. Spontaneous Intracranial Hypotension: A Systematic Imaging Approach for CSF Leak Localization and Management Based on MRI and Digital Subtraction Myelography. AJNR Am J Neuroradiol. 2019 Apr;40(4):745-753. doi: 10.3174/ajnr.A6016. Epub 2019 Mar 28. PMID 30923083
- [Background] Hani L, Fung C, El Rahal A, Volz F, Kraus LM, Schnell O, Ferrarese R, Erny D, Schwabenland M, Urbach H, Lutzen N, Beck J. Distinct Pattern of Membrane Formation With Spinal Cerebrospinal Fluid Leaks in Spontaneous Intracranial Hypotension. Oper Neurosurg. 2024 Jan 1;26(1):71-77. doi: 10.1227/ons.0000000000000914. Epub 2023 Sep 25. PMID 37747369
- [Background] Uppal V, Russell R, Sondekoppam RV, Ansari J, Baber Z, Chen Y, DelPizzo K, Dirzu DS, Kalagara H, Kissoon NR, Kranz PG, Leffert L, Lim G, Lobo C, Lucas DN, Moka E, Rodriguez SE, Sehmbi H, Vallejo MC, Volk T, Narouze S. Evidence-based clinical practice guidelines on postdural puncture headache: a consensus report from a multisociety international working group. Reg Anesth Pain Med. 2024 Jul 8;49(7):471-501. doi: 10.1136/rapm-2023-104817. PMID 37582578
- [Background] Jesse CM, Hani L, Fung C, Ulrich CT, Schar RT, Dobrocky T, Piechowiak EI, Goldberg J, Schankin C, Sintonen H, Beck J, Raabe A. The impact of spontaneous intracranial hypotension on social life and health-related quality of life. J Neurol. 2022 Oct;269(10):5466-5473. doi: 10.1007/s00415-022-11207-7. Epub 2022 Jun 14. PMID 35701531
- [Background] Beck J, Ulrich CT, Fung C, Fichtner J, Seidel K, Fiechter M, Hsieh K, Murek M, Bervini D, Meier N, Mono ML, Mordasini P, Hewer E, Z'Graggen WJ, Gralla J, Raabe A. Diskogenic microspurs as a major cause of intractable spontaneous intracranial hypotension. Neurology. 2016 Sep 20;87(12):1220-6. doi: 10.1212/WNL.0000000000003122. Epub 2016 Aug 26. PMID 27566748
- [Background] Kilic K, Korsbaek JJ, Jensen RH, Cvetkovic VV. Diagnosis of idiopathic intracranial hypertension - the importance of excluding secondary causes: A systematic review. Cephalalgia. 2022 May;42(6):524-541. doi: 10.1177/03331024211056580. Epub 2021 Nov 25. PMID 34822742
- [Background] Ducros A, Biousse V. Headache arising from idiopathic changes in CSF pressure. Lancet Neurol. 2015 Jun;14(6):655-68. doi: 10.1016/S1474-4422(15)00015-0. PMID 25987284
- [Background] Cheema S, Anderson J, Duncan C, Davagnanam I, Armstrong P, Redfern N, Ordman A, D'Antona L, Nissen J, Sayal P, Vaughan-Huxley E, Lagrata S, Iodice V, Snape-Burns J, Joy C, Matharu M. Survey of healthcare professionals' knowledge, attitudes and practices regarding spontaneous intracranial hypotension. BMJ Neurol Open. 2022 Sep 5;4(2):e000347. doi: 10.1136/bmjno-2022-000347. eCollection 2022. PMID 36110926
- [Background] Cheema S, Joy C, Pople J, Snape-Burns J, Trevarthen T, Matharu M. Patient experience of diagnosis and management of spontaneous intracranial hypotension: a cross-sectional online survey. BMJ Open. 2022 Jan 20;12(1):e057438. doi: 10.1136/bmjopen-2021-057438. PMID 35058269
- [Background] Hani L, Fung C, Jesse CM, Ulrich CT, Piechowiak EI, Gralla J, Raabe A, Dobrocky T, Beck J. Outcome after surgical treatment of cerebrospinal fluid leaks in spontaneous intracranial hypotension-a matter of time. J Neurol. 2022 Mar;269(3):1439-1446. doi: 10.1007/s00415-021-10710-7. Epub 2021 Jul 18. PMID 34274993
- [Background] Volz F, Fung C, Wolf K, Lutzen N, Urbach H, Kraus LM, Omer M, Beck J, El Rahal A. Recovery and long-term outcome after neurosurgical closure of spinal CSF leaks in patients with spontaneous intracranial hypotension. Cephalalgia. 2023 Aug;43(8):3331024231196808. doi: 10.1177/03331024231195830. PMID 37652456
- See also: Spinal CSF Leak Foundation - Home - Spinal CSF Leak Foundation. Accessed September 5, 2023 — https://spinalcsfleak.org/
- See also: Homepage. CSF Leak Association. Accessed September 5, 2023 — https://csfleak.uk/
- See also: SPINAL CSF LEAK CANADA. SPINAL CSF LEAK CANADA. Accessed September 5, 2023 — https://www.spinalcsfleakcanada.ca